## **Proposed Analyses**

Rates of procedure adherence (i.e., watching the video at least three times daily) will be assessed in order to examine the study's first question. The second question will be assessed by examining participants' rating of acceptability on the AARP with using a mobile phone as a method for self-directed exposure.

There will be 3 (group) x 2 (assessment) mixed measures analyses of variance (ANOVAs) which will be conducted to assess the first hypothesis regarding treatment effectiveness, with the DFS, and various DBAT measures (i.e., avoidance/escape, cardiac response, and SUDS verbal reports) as dependent variables. Sensitivity analyses will be conducted for baseline measurements. In order to examine the second hypothesis, a paired sample *t*-test assessing the relation of video perspective and scores on the PQ will be conducted.